CLINICAL TRIAL: NCT03833193
Title: Moderate Hypofractionated(3Gy/f) Radiotherapy for Advanced Lung Cancer: a Retrospective Study.
Brief Title: Moderate Hypofractionated Radiotherapy for Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: North China Petroleum Bureau General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NorthChinaPBGHA
Record Dates: First submitted 2019-02-03; First posted 2019-02-06 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Lung Cancer
Keywords: Hypofractionated radiotherapy;; Radiation-reduced esophagitis;; Radiation-reduced pneumonitis;Predictor
MeSH Terms: conditions — Lung Neoplasms | interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypofractionated radiotherapy (Experimental): The patients received daily accelerated radiotherapy with a total dose of 60Gy, delivered at 3Gy per fraction, five fractions per week, completed within 4 weeks.
  Interventions: Radiation: Hypofractionated radiotherapy

INTERVENTIONS:
Radiation: Hypofractionated radiotherapy — Radiation: Hypofractionated radiotherapy at 3Gy/f

SUMMARY:
The purpose of this study is to evaluate the incidences of Grade III and above radiation-reduced esophagitis and radiation-reduced pneumonia of patients with advanced lung cancer treated with moderate hypofractionated (3Gy/f) radiotherapy, and their predictors. Efficacies are also evaluated.

DETAILED DESCRIPTION:
Radiotherapy plays an irreplaceable role in lung cancer. However, due to the long duration of conventional fractionation irradiation, tumor cells will accelerate repopulation after 3 to 4 weeks during radiotherapy, resulting in decreased efficacy. Hypofractionated radiation is increasingly used in radiotherapy of lung cancer. It can shorten the overall treatment time, and can potentially reduce the effect of tumor accelerated repopulation. Compared with conventional radiotherapy, hypofractionated radiotherapy can theoretically obtain a higher biological effective dose (BED). The application of Stereotactic Body Radiation Therapy (SBRT) or Stereotactic Ablative Radiotherapy (SABR) in advanced or central lung cancer is restricted when the tumors are adjacent to important organs. Moderate hypofractionated radiotherapy can not only shorten the overall total treatment time, but also reduce the severe toxicities. It is widely used in lung cancer nowadays. However, most data of the tolerated doses for normal tissue and organs comes from conventional radiotherapy. Whether or not it is suitable for hypofractionated radiotherapy has not been determined. In our study, the incidences of Grade III and above radiation-reduced esophagitis and radiation-reduced pneumonia, as well as their predictors, were obtained by retrospective analysis of patients received moderate hypofractionated radiotherapy of 3Gy/f. At the same time, the efficacies of this scheme are also evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with previously untreated advanced lung cancer were recruited, who were confirmed pathologically or cytologically.
2. The Karnofsky performance status (KPS) score ≥60.
3. The expected survival time was≥3 months.
4. The laboratory examination results showed a neutrophil count ≥2.0 × 109, a hemoglobin level ≥100 g/L, a platelet count ≥100 × 109, and enough liver and kidney functions.
5. The patients did not show abnormal electrocardiogram (ECG) results.
6. They did not have other combined diseases that required hospitalization.
7. Informed consent required before enrollment.

Exclusion Criteria:

1. Patients who were pregnant or breastfeeding.
2. Patients who had another malignant tumor history (with the exception of patients with cervical carcinoma in situ and non-malignant melanoma skin cancer that had been clinically cured for at least 5 years), could not receive concurrent chemotherapy due to medical reasons.
3. Superior vena cava syndrome.
4. Syndrome and severe lung diseases that affected lung function were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade III and above radiation-reduced esophagitis | three years
  Incidence of grade III and above radiation-reduced esophagitis
Incidence of grade III and above radiation-reduced pneumonitis | three years
  Incidence of grade III and above radiation-reduced pneumonitis

SECONDARY OUTCOMES:
Objective Response Rate | three years
  ORR
Local Control Rate | three years
  LCR
Progression Free Survival | three years
  PFS
Median Survival Time | three years
  MST
Overall Survival | three years
  OS

CONTACTS AND LOCATIONS:
Overall Officials: QIANG LIN, Dr, Study Director — North China Petroleum Bureau General Hospital
Locations (1):
- North China Petroleum Bureau General Hospital, Cangzhou, Hebei, China

IPD SHARING:
Plan to Share IPD: No